CLINICAL TRIAL: NCT01886846
Title: Plasma Adiponectin Levels and Relations With Cytokines in Children With Acute Rheumatic Fever
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Dr Ali Yildirim, Fellow in Pediatric Cardiology, MD, Eskisehir Osmangazi University
Other Study IDs: EskisehirOU 4.6.2008/41
Record Dates: First submitted 2013-06-19; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Acute Rheumatic Fever
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

SUMMARY:
We aimed to investigate if adiponectin facilitates diagnosis of ARF by analyzing adiponectin levels in acute and convalescent periods of the acute rheumatic fever and by comparing results with that of healthy control group; also by comparatively examining levels of adiponectin in ARF cases who had different clinical findings at presentation. In addition, we aimed to investigate its role in the pathogenesis of ARF by evaluating correlations with cytokines such as TNF-α, IL-6 and IL-8 and acute phase reactants.

DETAILED DESCRIPTION:
Totally, 33 children (age range: 5 - 17 years; 15 male and 18 female) were enrolled to the study who were diagnosed as ARF at the Pediatric Cardiology Department, Medical Faculty, Eskişehir Osmangazi University. The study protocol was approved by Ethics Committee of Medical Faculty, Eskişehir Osmangazi University (Decision No. 41 dated June 4, 2008). Parents of study participants were informed about the aim and the method of the study and written consents were obtained.

For the study subjects, diagnosis of ARF was made according to the Modified Jones criteria (4) and appropriate treatment was started. Patients were divided into three groups by clinical findings. Group 1 included patients with only chorea, while patients with arthritis and carditis were involved in Group 2 and patients with only carditis were included in the Group 3. A group with only arthritis was not established since the patients with isolated arthritis are usually followed up at primary and secondary healthcare facilities rather than referring those patients to our tertiary healthcare center.

Venous Blood Sampling Following tests were analyzed using venous blood samples drawn from patients and healthy control subjects; complete blood count, ESR, nephelometric CRP and immune turbidimetric hsCRP, total cholesterol, triglyceride, LDL-C and HDL-C levels by enzymatic coloxrimetric method and FSH and LH and total testosterone (for male subjects) and estradiol (for female subjects)levels by chemoluminescent assey. Plasma and serum samples were drawn for adiponectin, TNF-α, IL-6 and IL-8. Blood samples were drawn for analyzing acute phase reactants at Day 2nd , 5th , 10th and 15th days and at 8 week in order to evaluate response to the treatment, while blood samples were simultaneously drawn for analyzing adiponectin, TNF-α, IL-6 and IL-8 levels.

Plasma Adiponectin Measurement Venous blood samples were added into the centrifuge tubes with EDTA, they were centrifuged at 3000 rpm, 4 °C for 15 minutes and the resultant plasma samples were stored at -80 °C. Plasma samples were diluted (1:300) as directed by the instruction for use of the kit, before the analysis was conducted. Samples taken for plasma adiponectin levels were analyzed using Human Adiponectin ELISA, High Sensitivity kit (BioVendor Research and Diagnostic Products, Modrice, Czech Republic) with enzyme-linked immunosorbent assay (ELISA) method. Absorbance was read at 450 nm. Results were expressed as ng/ml and converted into µg/ml via dividing them by 1000.

Serum TNF-α, IL-6 and IL-8 Measurements The venous blood samples were added into centrifuge tubes not containing anticoagulant for measuring serum TNF-α, IL-6 and IL-8 levels. Samples were centrifuged at 3000 rpm, 4 °C for 15 minutes and the resultant serum samples were stored at -80 °C. Samples taken for measuring serum TNF-, IL-6 and IL-8 levels were analyzed with ELISA method using Human TNF-α ELISA, Human IL-6 ELISA, Human IL-8/NAP-1 ELISA kits (Bender MedSystems, Vienna, Austria). Absorbance was read at 450 nm. Results were expressed as pg/ml.

ELIGIBILITY:
For the study subjects, diagnosis of ARF was made according to the Modified Jones criteria (4) and appropriate treatment was started. Patients were divided into three groups by clinical findings. Group 1 included patients with only chorea, while patients with arthritis and carditis were involved in Group 2 and patients with only carditis were included in the Group 3. A group with only arthritis was not established since the patients with isolated arthritis are usually followed up at primary and secondary healthcare facilities rather than referring those patients to our tertiary healthcare center.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: acute rheumatic fever and by comparing results with that of healthy
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline adiponectin and cytokin levels at 2 months in the acute rheumatic fever | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi Universty, Eskişehir, Odunpazarı, Turkey (Türkiye)

REFERENCES:
- [Background] Ouchi N, Walsh K. Adiponectin as an anti-inflammatory factor. Clin Chim Acta. 2007 May 1;380(1-2):24-30. doi: 10.1016/j.cca.2007.01.026. Epub 2007 Feb 2. PMID 17343838